CLINICAL TRIAL: NCT03990636
Title: Photodynamic Therapy With Metil 5-aminolevulinate for Actinic Cheilitis - A Phase 2 Randomized Double-blind Placebo Controlled Clinical Trial
Brief Title: Photodynamic Therapy With Metil 5-aminolevulinate for Actinic Cheilitis - Phase 2 Clinical Trial
Acronym: PDTMALAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Daniel Cohen Goldenberg, Photodynamic therapy with methyl aminolevulinate in the treatment of actinic cheilitis, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCABrazilCOPQ
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Actinic Cheilitis; Leukoplakia; Erythroplakia
Keywords: PDT; Actinic Cheilitis; Phase 2 Clinical Trial
MeSH Terms: conditions — Actinic cheilitis; Leukoplakia; Erythroplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metil 5-aminolevulinate arm (Experimental): Metil 5-aminolevulinate arm with photo activation.
  Interventions: Drug: Metil 5-aminolevulinate
- Placebo arm (Placebo Comparator): Placebo (without metil 5-aminolevulinate) arm with photo activation.
  Interventions: Drug: Metil 5-aminolevulinate

INTERVENTIONS:
Drug: Metil 5-aminolevulinate — Scrubbing lip vermillion and applying the medication or placebo that is activated (or not, in case of placebo) with red light.

SUMMARY:
Brazil is a tropical country, with high incidence of ultraviolet radiation throughout the year. Many Europeans migrated to Brazil escaping either war or economic crisis to live in the country searching for opportunities. Low phototype combined with high incidence of UV light is a combination that not only affect the skin but also the lips. The current study was designed to use photodynamic therapy with metil 5-aminolevulinate for actinic cheilitis in a phase 2 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis with histopathological confirmation of actinic cheilitis
* Patients will be requested to respect the timeframe of clinical consultations
* No treatment for actinic cheilitis in the last 3 months

Exclusion Criteria:

* Histopathological diagnosis of squamous cell carcinoma (SCC)
* Patient presenting any type of immunosupression
* Recurrent crust of the lip vermilion (high risk of SCC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-17 (Estimated); Primary Completion 2020-05-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response | 18 months
  Expected complete clinical response in 60% of cases
Histological cure | 18 months
  Expected histological cure in 40% of cases

SECONDARY OUTCOMES:
IHC analysis | 18 months
  Expression of immunohistochemical markers of cancer progression

IPD SHARING:
Plan to Share IPD: No
The Informed Consent Form (ICF) will be read and explained to each patient informing about all the risks and potential benefits. Clinical Study Report (CSR) is going to be registered for all patients, although data will not be shared.